CLINICAL TRIAL: NCT02871232
Title: Extended-Release (ER) and Long-Acting (LA) Opioid Analgesics Risk Evaluation and Mitigation Strategy (REMS): RADARS® System Surveillance Protocol
Brief Title: Surveillance Monitoring of Opioid Abuse in Poison and Drug Treatment Centers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ER/LA Opioid REMS Program Companies (RPC) (Industry)
Responsible Party: Sponsor
Other Study IDs: Assessments 5.2-5.4
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Opioid-related Disorders; Opioid Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (2):
- Intentional exposures among adolescents and adults
  Interventions: Other: Researched Abuse, Diversion and Addiction-Related Surveillance (RADARS) System of post-marketing surveillance of prescription medication abuse, misuse, and diversion
- Unintentional exposures among infants and children
  Interventions: Other: Researched Abuse, Diversion and Addiction-Related Surveillance (RADARS) System of post-marketing surveillance of prescription medication abuse, misuse, and diversion

INTERVENTIONS:
Other: Researched Abuse, Diversion and Addiction-Related Surveillance (RADARS) System of post-marketing surveillance of prescription medication abuse, misuse, and diversion

SUMMARY:
To conduct surveillance for abuse, misuse, overdose, addiction, and death and to evaluate if the REMS meets its surveillance goals, and if it does not, to modify it appropriately based on the metrics. Briefly, therefore, the overall surveillance objective is to evaluate for trends before and after the shared REMS is implemented to collectively assess for changes in abuse, misuse, overdose, addiction, and death for different risk groups and settings.

ELIGIBILITY:
Inclusion Criteria:

Any patient with data in the RADARS system

Exclusion Criteria:

None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The Poison Center Program obtains data from the general population of the US, Treatment Center Programs obtain data from those entering treatment for opioid addiction, and the College Survey Program surveys self-identified students attending a 2- or 4- year college, university, or technical school
Sampling Method: Non-Probability Sample
Enrollment: 26500 (Estimated)
Dates: Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Poisson regression will be used to compare changes in rates of abuse, misuse, overdose, and death and other outcomes over time within the ER/LA opioid group to changes in rates among the comparator groups | Review over period from January 2010 to December 2016

SECONDARY OUTCOMES:
Mean number of dosing units per prescriptions dispensed across time for the ER/LA REMS drug group | Review over period from January 2010 to December 2016